CLINICAL TRIAL: NCT01708278
Title: Phase I Study to Determine the Safety of Quercetin in COPD Patients
Brief Title: Beneficial Effects of Quercetin in Chronic Obstructive Pulmonary Disease (COPD)
Acronym: Quercetin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Institutes of Health (NIH) (NIH); Quercegen Pharmaceuticals (Industry); National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Umadevi S. Sajjan, Assistant Professor, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HUM00061735; R21AT007357 (NIH); NCT02013440 (obsolete NCT alias)
Record Dates: First submitted 2012-10-10; First posted 2012-10-16 (Estimated); Results first posted 2016-12-26 (Estimated); Last update posted 2016-12-26 (Estimated); Status verified 2016-10

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD; Emphysema; chronic bronchitis; Quercetin; flavonoids
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Emphysema; Bronchitis, Chronic | interventions — Quercetin; Folic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Sugar chew-Cohort 1 (Placebo Comparator): contains 350 mg of vitamin C and 10 mg niacin
  Interventions: Other: Placebo - sugar chew
- Quercetin 1-Cohort 1 (Active Comparator): Quercetin chew containing 500 mg quercetin, 350 mg vitamin C and 10 mg niacin
  Interventions: Drug: Quercetin
- Quercetin 2-Cohort 2 (Active Comparator): Quercetin chew containing 1000 mg quercetin, 350 mg vitamin C and 10 mg niacin
  Interventions: Drug: Quercetin
- Quercetin 3-Cohort 3 (Active Comparator): Quercetin chew containing 2000 mg quercetin, 350 mg vitamin C and 10 mg niacin
  Interventions: Drug: Quercetin
- Sugar chew-Cohort 2 (Placebo Comparator): contains 350 mg of vitamin C and 10 mg niacin
  Interventions: Other: Placebo - sugar chew
- Sugar Chew-Cohort 3 (Placebo Comparator): contains 350 mg of vitamin C and 10 mg niacin
  Interventions: Other: Placebo - sugar chew

INTERVENTIONS:
Drug: Quercetin — COPD Subjects will be asked to avoid quercetin rich diet for one week and then asked to take one of the following for 1 week
  1. Quercetin 500 mg/350 mg of vitamin C and 10 mg niacin
  2. Quercetin 1000 mg/350 mg of vitamin C and 10 mg niacin
  3. Quercetin 2000 mg/350 mg of vitamin C and 10 mg niacin
  Other Names: QB3C without folic acid
  Arms: Quercetin 1-Cohort 1; Quercetin 2-Cohort 2; Quercetin 3-Cohort 3
Other: Placebo - sugar chew — COPD Subjects will be asked to avoid quercetin rich diet for one week and then asked to take placebo (sugar chew containing 350 mg of vitamin C and 10 mg niacin)
  Arms: Sugar Chew-Cohort 3; Sugar chew-Cohort 1; Sugar chew-Cohort 2

SUMMARY:
Chronic obstructive pulmonary disease (COPD) is a progressive disorder of the lung parenchyma and airways, which is the third-leading cause of death in the USA. Current therapies for COPD are only partially effective and may also have side effects. Although increasing evidence indicates that quercetin supplementation may be beneficial in treating COPD, key methodological issues have not been resolved. The overall objective of this study is to determine the dosage of quercetin supplementation, bioavailability of quercetin, safety, dose-response relationship and appropriate biomarkers which reflect clinical outcomes in patients with COPD that is necessary for conducting large clinical trials in this patient population.

DETAILED DESCRIPTION:
In our preclinical study, we have demonstrated that 4 fold increase in plasma quercetin levels significantly decreased lung inflammation and prevented progression. Clinical studies in healthy volunteers 4 fold increase in plasma quercetin levels (0.22 to 1 µM) could be achieved by supplementing with 500mg of quercetin/day. However, safety of quercetin supplementation and quercetin dose required to achieve 4 fold increases in plasma quercetin levels in 'at-high-risk' COPD population is yet to be established. This study involves two phases; the first phase examines the safety of quercetin supplementation in subjects with chronic obstructive pulmonary disease (COPD) and the second phase determines the efficacy of quercetin in COPD patients. In this study, we will enroll COPD patients with mild to moderate disease between the age group of 40 to 65 years. During the first phase, we will enroll a total of 9 patients to examine the tolerance and safety of three doses of quercetin (500, 1000 and 2000 mg/day) in a dose escalation manner. First cohort consisting of three subjects will receive placebo or 500 mg of quercetin per day for one week and the safety of quercetin supplementation will be assessed by monitoring adverse events and any changes in outcomes of blood test that include complete blood counts (CBC)and comprehensive metabolic panel prior to after supplementation. If this dose is safe and tolerated, second cohort of 3 subjects will receive placebo or 1000 mg of quercetin per day quercetin for one week and again safety will be assessed. If the dose is safely tolerated, the third cohort will receive either placebo or 2000 mg of quercetin per day for a week and the safety will be assessed.

Having completed Phase I study at University of Michigan, we planned to do the Phase II efficacy study under separate NCT number. As of 2016 this phase II study has not begun. Based on the initial study, we plan to choose the highest quercetin dose tolerated with no adverse events and the dose (500 mg of quercetin per day) that was found to increase plasma quercetin levels by 4 fold over baseline in healthy volunteers to examine the efficacy of quercetin in reducing inflammatory and oxidative stress markers and improving lung function in COPD subjects. In the second phase, we will enroll a total of 75 subjects and randomized into three arms; placebo (15 subjects) or one of the two doses of quercetin (30 subjects per arm). All enrolled subjects will be asked to avoid quercetin rich foods throughout the study period. One week after enrollment (run-in), subjects will be either supplemented with either placebo or one of the two doses of quercetin for 4 weeks. All participants will be blinded for study agents. Plasma and sputum quercetin levels, lung function, and markers of oxidative stress and inflammation will be determined at the start of the study (following run-in period), at the end of 4 weeks treatment period.

Three of the original outcome measures listed related to this follow up study of 4 weeks treatment which was never begun. Therefore they have been deleted.

ELIGIBILITY:
Inclusion Criteria:

* Subjects diagnosed with mild to moderate COPD (GOLD stage I, II and III)-
* 10 pack-year smoking history or greater and ceased to smoke at least for 2 months prior to recruitment
* Subjects taking H2 antagonists, Imodium or loratadine and willing to stop during the study period

Exclusion criteria:

* COPD subjects with >80% or <35% predicted
* Current smokers
* Known allergy/sensitivity to quercetin
* Subjects with primary diagnosis of asthma
* Upper respiratory tract infection within two weeks of the screening visit
* Acute bacterial infection requiring antibiotics within two weeks of screening
* Emergency treatment or hospitalization within one month of screening
* Pregnant or lactating mothers
* Women who don't consent to take pregnancy test
* Unwillingness to stop flavonoid supplementation
* Dietary intake exceeding or averaging 150 mg quercetin daily as assessed by Bioflavonoid Food and Supplement Screener
* Daily oral steroid treatment, warfarin, cyclosporine (neural, sandimmune), digoxin, fexofenadine, paclitaxel, diltiazem, saquinavir, selected chemotherapeutic agents (etoposide, vinblastine, vincristine, vindesine), antifungals (ketoconazole, itraconazole), protease inhibitors (amprenavir, indinavir, nelfinavir), verapamil, oral glucocorticoids, erythromycin, quinidine
* Subjects taking H2 antagonists (cimetidine, ranitidine), loperamide (Imodium) or loratadine and not willing to stop during study period
* Lung cancer history or undergoing chemo- or radiation therapy
* Inflammatory bowel disease
* Child bearing age, who are unwilling to use adequate contraception or abstain during the course of the study.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2014-02; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Fernando J Martinez, M.D., Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

REFERENCES:
- [Background] Ganesan S, Faris AN, Comstock AT, Chattoraj SS, Chattoraj A, Burgess JR, Curtis JL, Martinez FJ, Zick S, Hershenson MB, Sajjan US. Quercetin prevents progression of disease in elastase/LPS-exposed mice by negatively regulating MMP expression. Respir Res. 2010 Sep 28;11(1):131. doi: 10.1186/1465-9921-11-131. PMID 20920189
- [Background] Ganesan S, Faris AN, Comstock AT, Wang Q, Nanua S, Hershenson MB, Sajjan US. Quercetin inhibits rhinovirus replication in vitro and in vivo. Antiviral Res. 2012 Jun;94(3):258-71. doi: 10.1016/j.antiviral.2012.03.005. Epub 2012 Mar 23. PMID 22465313
- [Background] Comstock AT, Ganesan S, Chattoraj A, Faris AN, Margolis BL, Hershenson MB, Sajjan US. Rhinovirus-induced barrier dysfunction in polarized airway epithelial cells is mediated by NADPH oxidase 1. J Virol. 2011 Jul;85(13):6795-808. doi: 10.1128/JVI.02074-10. Epub 2011 Apr 20. PMID 21507984
- [Background] Jin F, Nieman DC, Shanely RA, Knab AM, Austin MD, Sha W. The variable plasma quercetin response to 12-week quercetin supplementation in humans. Eur J Clin Nutr. 2010 Jul;64(7):692-7. doi: 10.1038/ejcn.2010.91. Epub 2010 Jun 2. PMID 20517329
- [Background] Boots AW, Wilms LC, Swennen EL, Kleinjans JC, Bast A, Haenen GR. In vitro and ex vivo anti-inflammatory activity of quercetin in healthy volunteers. Nutrition. 2008 Jul-Aug;24(7-8):703-10. doi: 10.1016/j.nut.2008.03.023. PMID 18549926
- [Background] Terao J, Murota K, Kawai Y. Conjugated quercetin glucuronides as bioactive metabolites and precursors of aglycone in vivo. Food Funct. 2011 Jan;2(1):11-7. doi: 10.1039/c0fo00106f. Epub 2010 Nov 17. PMID 21773581
- [Background] Boots AW, Drent M, de Boer VC, Bast A, Haenen GR. Quercetin reduces markers of oxidative stress and inflammation in sarcoidosis. Clin Nutr. 2011 Aug;30(4):506-12. doi: 10.1016/j.clnu.2011.01.010. Epub 2011 Feb 15. PMID 21324570
- [Background] Bischoff SC. Quercetin: potentials in the prevention and therapy of disease. Curr Opin Clin Nutr Metab Care. 2008 Nov;11(6):733-40. doi: 10.1097/MCO.0b013e32831394b8. PMID 18827577
- [Background] Harwood M, Danielewska-Nikiel B, Borzelleca JF, Flamm GW, Williams GM, Lines TC. A critical review of the data related to the safety of quercetin and lack of evidence of in vivo toxicity, including lack of genotoxic/carcinogenic properties. Food Chem Toxicol. 2007 Nov;45(11):2179-205. doi: 10.1016/j.fct.2007.05.015. Epub 2007 Jun 7. PMID 17698276
- [Background] Okamoto T. Safety of quercetin for clinical application (Review). Int J Mol Med. 2005 Aug;16(2):275-8. PMID 16012761
- [Derived] Han MK, Barreto TA, Martinez FJ, Comstock AT, Sajjan US. Randomised clinical trial to determine the safety of quercetin supplementation in patients with chronic obstructive pulmonary disease. BMJ Open Respir Res. 2020 Feb;7(1):e000392. doi: 10.1136/bmjresp-2018-000392. PMID 32071149

RESULTS

PARTICIPANT FLOW:
Groups:
- Sugar Chew- Cohort 1; Sugar Chew-Cohort 2; Sugar Chew-Cohort 3: contains 350 mg of vitamin C and 10 mg niacin
  Placebo - sugar chew: COPD Subjects will be asked to avoid quercetin rich diet for one week and then asked to take placebo (sugar chew containing 350 mg of vitamin C and 10 mg niacin)
- Quercetin 1-Cohort 1: Quercetin chew containing 500 mg quercetin, 350 mg vitamin C and 10 mg niacin
  Quercetin: COPD Subjects will be asked to avoid quercetin rich diet for one week and then asked to take one of the following for 1 week
  1. Quercetin 500 mg/350 mg of vitamin C and 10 mg niacin
  2. Quercetin 1000 mg/350 mg of vitamin C and 10 mg niacin
  3. Quercetin 2000 mg/350 mg of vitamin C and 10 mg niacin
- Quercetin 2-Cohort 2: Quercetin chew containing 1000 mg quercetin, 350 mg vitamin C and 10 mg niacin
  Quercetin: COPD Subjects will be asked to avoid quercetin rich diet for one week and then asked to take one of the following for 1 week
  1. Quercetin 500 mg/350 mg of vitamin C and 10 mg niacin
  2. Quercetin 1000 mg/350 mg of vitamin C and 10 mg niacin
  3. Quercetin 2000 mg/350 mg of vitamin C and 10 mg niacin
- Quercetin 3-Cohort 3: Quercetin chew containing 2000 mg quercetin, 350 mg vitamin C and 10 mg niacin
  Quercetin: COPD Subjects will be asked to avoid quercetin rich diet for one week and then asked to take one of the following for 1 week
  1. Quercetin 500 mg/350 mg of vitamin C and 10 mg niacin
  2. Quercetin 1000 mg/350 mg of vitamin C and 10 mg niacin
  3. Quercetin 2000 mg/350 mg of vitamin C and 10 mg niacin
Period: Overall Study
Arm/Group | Sugar Chew- Cohort 1 | Quercetin 1-Cohort 1 | Quercetin 2-Cohort 2 | Quercetin 3-Cohort 3 | Sugar Chew-Cohort 2 | Sugar Chew-Cohort 3
Started | 1 | 2 | 2 | 2 | 1 | 1
Completed | 1 | 2 | 2 | 2 | 1 | 1
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sugar Chew- Cohort 1 | Quercetin 1-Cohort 1 | Quercetin 2-Cohort 2 | Quercetin 3-Cohort 3 | Sugar Chew-Cohort 2 | Sugar Chew-Cohort 3 | Total
Number analyzed (Participants) | 1 | 2 | 2 | 2 | 1 | 1 | 9
Age, Customized [Number; unit: participants]
  Age 40 - 80 years | 1 | 2 | 2 | 2 | 1 | 1 | 9
Gender [Count of Participants; unit: Participants]
  Female | 1 | 1 | 0 | 1 | 1 | 0 | 4
  Male | 0 | 1 | 2 | 1 | 0 | 1 | 5
Region of Enrollment [Number; unit: participants]
  United States | 1 | 2 | 2 | 2 | 1 | 1 | 9
Lung Function [Number; unit: participants] — Lung Function FEV1 between 35 and 80% predicted
  participants | 1 | 2 | 2 | 2 | 1 | 1 | 9

OUTCOME MEASURES:

1. Primary Outcome: Participants Who Experienced Safety Concerns, Where Safety Concerns of Quercetin Supplementation is Indicated by Significant Change From Baseline Measures of Tests Indicated Below in Outcome Measure Description
Description: Note: If values for any of the measures indicated here were found, the participant would be indicated as a participant with a safety concern, and values for that particular measure would be posted specifically, but since none of the participants experienced these outlying values, results of all tests are expressed here as a composite function.
  PULMONARY FUNCTION TEST:
  FEV1% of predicted: decline by >20% from baseline COMPLETE BLOOD COUNTS: WBC (cells)/mm3 : <2000, Platelets (cells)/mm3: <25,000, Hemoglobin (g/dL): <7.0 COMPREHENSIVE METABOLIC PROFILE (study drug related):Sodium (mmol/L): <125 or >148, Potassium (mmol/L): < 3.0 or > 6.0, Calcium (mmol/L): <7.4 or > 11.5, LIVER FUNCTION TESTS INCREASE BY FACTOR: Enzymes ALT, AST, and Alkaline phosphate, Total bilirubin: for any of these a value >3X upper limit of normal
Time Frame: One week in Phase I safety study
Measure: Count of Participants; unit: Participants
Arm/Group | Sugar Chew- Cohort 1 | Quercetin 1-Cohort 1 | Quercetin 2-Cohort 2 | Quercetin 3-Cohort 3 | Sugar Chew-Cohort 2 | Sugar Chew-Cohort 3
Number analyzed (Participants) | 1 | 2 | 2 | 2 | 1 | 1
Participants | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: 14 days
Arm/Group | Sugar Chew-Cohort 1 | Quercetin 1-Cohort 1 | Quercetin 2-Cohort 2 | Quercetin 3-Cohort 3 | Sugar Chew-Cohort 2 | Sugar Chew-Cohort 3
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/2 | 0/2 | 0/2 | 0/1 | 0/1
Other Adverse Events (participants affected / at risk) | 1/1 | 2/2 | 2/2 | 1/2 | 1/1 | 1/1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Sugar Chew-Cohort 1 (N=1) | Quercetin 1-Cohort 1 (N=2) | Quercetin 2-Cohort 2 (N=2) | Quercetin 3-Cohort 3 (N=2) | Sugar Chew-Cohort 2 (N=1) | Sugar Chew-Cohort 3 (N=1)
Heart burn, GERD (Gastrointestinal disorders) | 1 | 1 | 1 | 0 | 0/0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Congestion/Breathlessness/chest tightness/cough (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 1 | 1 | 1 | 1
Sleep disturbance (Nervous system disorders) | 1 | 1 | 1 | 0 | 1 | 1
headache/neck pain/low back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0
high glucose (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0
Flu (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes